CLINICAL TRIAL: NCT04480190
Title: Feasibility of Total Neoadjuvant Therapy in Resectable Biliary Adenocarcinoma
Brief Title: Neoadjuvant Therapy in Biliary Adenocarcinoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Difficulty accruing
Sponsor: Jordan Kharofa (Other)
Responsible Party: Sponsor-Investigator, Jordan Kharofa, Principal Investigator, University of Cincinnati
Organization: University of Cincinnati (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCCC-GI-20-01
Record Dates: First submitted 2020-06-25; First posted 2020-07-21 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Cholangiocarcinoma; Biliary Cancer
MeSH Terms: conditions — Cholangiocarcinoma; Biliary Tract Neoplasms | interventions — Gemcitabine; Cisplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- Research Treatment (Experimental): Gemcitabine/Cisplatin/ChemoRT
  Interventions: Drug: Gemcitabine; Drug: Cisplatin; Drug: Fluorouracil; Radiation: Short course ChemoRT

INTERVENTIONS:
Drug: Gemcitabine — IV Gemcitabine 1000mg/m2 to be given on Days 1, Day 8 (Before Cisplatin); 3 week cycles
  Other Names: Gemzar
Drug: Cisplatin — IV Cisplatin 25mg/m2 to be given on Days 1, Day 8
  Other Names: Platinol
Drug: Fluorouracil — Infusional 5-FU 225 mg/m2/d via Continuous IV infusion, to be given Days 1-5 and 8-12 during RT
  Other Names: 5FU
Radiation: Short course ChemoRT — Radiation Therapy:
  Sim: All patients will undergo 4D-CT simulation with 3 hours fasting with or without IV contrast. Compression may be used depending on the tumor motion.
  Radiation Target Volume: The gross tumor volume (GTV) will be defined on all relevant imaging datasets including diagnostic CT, MRI, MRCP and/or ERCP data. An iGTV will be generated using the 4D datasets. The clinical target volume (CTV) will include the entire iGTV as well as portal lymphatic and celiac nodal space for all patients with selective treatment of the SMA and pancreaticoduodenal depending on the tumor location. A 5 mm margin will be added to the CTV to generate the planning target volume (PTV).
  Radiation Dose: The dose will be 30 Gy in 10 fractions (3 Gy per fraction) for all patients using either 3D Conformal or Intensity Modulated Radiation Therapy techniques.
  Other Names: ChemoRT

SUMMARY:
Feasibility of neoadjuvant therapy in resectable biliary adenocarcinoma.

DETAILED DESCRIPTION:
This trial will evaluate whether a neoadjuvant paradigm is feasible in resectable biliary adenocarcinoma. All components of therapy are currently used standards of care, however they have not been used in the neoadjuvant setting for the management of resectable biliary cancers. The study will use Gemcitabine/cisplatin, followed by chemoradiation.

This is a feasibility trial with an accrual goal of 12 patients using the primary endpoint of completion of neoadjuvant therapy and surgery as an assessment of feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* ECOG performance status ≤2
* Patients must have adequate organ and marrow function as defined below:

leukocytes ≥3,000/mcL absolute neutrophil count ≥1,500/mcL platelets ≥100,000/mcL total bilirubin ≤ 7 AST(SGOT)/ALT(SGPT) ≤3 × institutional ULN creatinine ≤ institutional ULN OR glomerular filtration rate (GFR) ≥ 30 mL/min/1.73 m2

* Known human immunodeficiency virus (HIV)-infected patients must be on effective anti-retroviral therapy with undetectable viral load within 6 months to be eligible for this trial.
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated.
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better.
* Patients must have either biopsy proven biliary adenocarcinoma (Intrahepatic cholangiocarcinoma, hilar cholangiocarcinoma, extrahepatic cholangiocarcinoma), or Gallbladder Adenocarcinoma or cytology with FISH abnormality sufficient for diagnosis.
* Patients must be deemed to have tumor that is resectable by the surgical oncologist and must have no medical contraindications to surgery.
* All patients must have a CT scan of the chest, abdomen, and pelvis with contrast or PET scan demonstrating no evidence of metastatic disease within 6 weeks prior to protocol therapy.
* Patients with enlarged regional lymph nodes within the dissection basin are eligible for participation.
* Women of child-bearing potential and men must agree to use adequate contraception for 14 months (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 14 months after completion.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients with metastatic disease on imaging (biopsy not required).
* Patients not eligible for surgery due to tumor anatomy or medical comorbidities.
* Patients with known hypersensitivity to cisplatin, gemcitabine or 5-FU or any component of the formulation.
* Patients who have had chemotherapy or radiotherapy within 3 months prior to entering the study.
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > Grade 1) with the exception of alopecia.
* Patients who are currently receiving any other investigational agents are excluded. Patients who received investigational agents prior to consenting to participate on this study who are no longer currently receiving those agents, are eligible.
* Patients with uncontrolled intercurrent illness that would prevent receipt of standard of care chemotherapy, radiation or surgery.
* Patients with psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02-04 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
Completion of all therapy. Defined as completing 4/6 doses of gem/cis chemo, 80% of RT dose, and surgical resection. | 5 years
  Feasibility trial with accrual goal of 12 patients using primary endpoint of completion of neoadjuvant therapy and surgery as an assessment of feasibility. Interim assessment of first 6 patients enrolled will be performed. Resection rate benchmark for neoadjuvant pancreas trials ~70% accounting for patients found to have progression. Completion of all therapy is defined as completing 4/6 doses of gem/cis chemo, 80% of RT dose, and surgical resection. If 2 or less of first 6 patients enrolled complete all therapy the trial will be closed and treatment will be considered unfeasible. Upon trial completion, if 5 or less of 12 patients complete all therapy the trial will be deemed unfeasible.

SECONDARY OUTCOMES:
Patients will be evaluated for toxicity during protocol therapy and postoperatively using the CTCAE v 5 criteria. | 5 years
  All patients will be evaluable for toxicity from the time of their first treatment with Gemcitabine/cisplatin using the CTCAE v 5 criteria.
Margin negative resection rate. This will be measured by the Proportion of patients with involved surgical margins (R1 rate). | 5 years
  This is one of the Pathologic outcomes that will be measured. The margin negative resection rate will be measured by the Proportion of patients with involved surgical margins (R1 rate).
Lymph node involvement. This will be measured by the Proportion of patients with involved lymph nodes (N0 vs N1). | 5 years
  This is one of the Pathologic outcomes that will be measured. Lymph node involvement will be measured by the Proportion of patients with involved lymph nodes (N0 vs N1).
Survival outcomes measured by Disease Free Survival [DFS]) | 5 years
  Disease-free survival: From date of registration to date of first documentation of relapse or death due to any cause. Patients last known to be alive and free of disease will be censored at date of last contact.
Survival outcomes measured by Local Failure Free Survival [LFFS]. | 5 years
  Local failure free survival: From date of registration to date of first documentation of local relapse or death due to any cause. Patients last known to be alive and without evidence of local relapse will be censored at date of last contact.
  Local relapse: Any evidence of new disease within the primary tumor bed or the regional (retroperitoneal, celiac, and portal vein nodes) lymphatics (these areas are to be encompassed within the radiation fields).
Survival outcomes measured by Overall Survival [OS]. | 5 years
  Overall Survival: From date of registration to date of death due to any cause. Patients last known to be alive will be censored at date of last contact.

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Kharofa, MD, Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No